CLINICAL TRIAL: NCT03767712
Title: Trauma as a Trigger for Autoimmunity - a Single Centre Observational Cohort Study
Brief Title: Trauma as a Trigger for Autoimmunity
Acronym: TATA
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-00895, me16Potlukova
Record Dates: First submitted 2018-12-04; First posted 2018-12-07 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Autoimmunity
Keywords: trauma; immunological reaction to trauma; pertrochanteric femoral fracture; antinuclear antibodies; activation of innate immunity; adaptive immunity
MeSH Terms: conditions — Autoimmune Diseases; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum samples of each subject in a form of biobank (TATA-Biobank) in order to allow future analyses (e.g. emerging biomarkers in relation to trauma).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Comparison of the levels of antinuclear antibodies (ANA) by indirect immunofluorescence on a Hep-2 cell line. — To analyse whether patients with pertrochanteric femoral fracture with consecutive gamma-nailing develop any laboratory signs of transient autoimmunity (comparison of the levels of ANA; in order to overcome the problem of subjective semiquantitative evaluation, the novel method of automated digital fluorescence microscopy will be used)

SUMMARY:
To analyse the immunological reaction to Trauma (pertrochanteric femoral fracture with consequent osteosynthesis) in the first weeks up to one year postoperatively with focus on the development of autoimmunity.

DETAILED DESCRIPTION:
This project represents a unique study of the influence of trauma on the immune system. It addresses the question whether an excess of apoptotic/necrotic cells can induce an at least transient autoimmune phenomena in humans. If the hypothesis of a transient induction of autoimmunity by trauma proves to be correct, this study will provide a novel insight into the pathogenesis of autoimmune diseases.

ELIGIBILITY:
Inclusion Criteria:

* pertrochanteric femoral fracture (≤7 days)
* planned gamma nail osteosynthesis
* ability to give written informed consent

Exclusion Criteria:

* Severe hepatic and renal failure
* current active oncological disease
* current immunosuppressive or biological therapy
* known systemic autoimmune disease
* foreseeable lack of complete follow-up (e.g. due to generally poor health)
* cognitive impairment (delirium, dementia, alteration of consciousness)
* insufficient knowledge of project language
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute pertrochanteric fracture in whom an operation (gamma-nail osteosynthesis) is planned at the University Hospital Basel.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-07-04 (Actual); Primary Completion 2019-12-23 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Change in ANA | Preoperative (1-2 days preoperative) and 12 weeks postoperative
  Fluorescence Index (FI) for ANA measurement (automated digital fluorescence microscopy = indirect immunofluorescence on a Hep-2 cell line). In order to overcome the problem of subjective semiquantitative evaluation, the novel method of automated digital fluorescence microscopy will be used (NOVA View, INOVA Diagnostics

SECONDARY OUTCOMES:
Change in ANA | 6 weeks postoperative and 12 weeks postoperative and 12 months postoperative
  Fluorescence Index (FI) for ANA measurement (automated digital fluorescence microscopy)
Change in Antibody level against double stranded deoxyribonucleic acid (Anti-dsDNA) | Preoperative (1-2 days preoperative) and 6 weeks postoperative and 12 weeks postoperative and 12 months postoperative
  serum level of Anti-dsDNA (U/ml)
Change in Antibody level against Anti-Cardiolipin | Preoperative (1-2 days preoperative) and 6 weeks postoperative and 12 weeks postoperative and 12 months postoperative
  serum level of Anti-Cardiolipin (U/ml)
Change in Antibody level against complement component C1q (Anti-C1q) | Preoperative (1-2 days preoperative) and 6 weeks postoperative and 12 weeks postoperative and 12 months postoperative
  serum level of C1q (U/ml)
Change in Antibody level against Sjögren's-syndrome-related antigen A (Anti-SSA/Ro) | Preoperative (1-2 days preoperative) and 6 weeks postoperative and 12 weeks postoperative and 12 months postoperative
  serum level of Anti-SSA/Ro (U/ml)
Change in proportion of immune cells (Plasmablasts, regulatory T cell (T-regs), total Cluster of Differentiation (CD)4+, CD8+, CD19+, Natural killer (NK) cells | Preoperative (1-2 days preoperative) and 3-4 days postoperative and 6 weeks postoperative and 12 weeks postoperative
  Change in proportion of immune cells (Plasmablasts, regulatory T cell (T-regs), total Cluster of Differentiation (CD)4+, CD8+, CD19+, Natural killer (NK) cells (cells/ml)
Change in serum levels of cytokines (Interleukin (IL)-6 , IL-10, IL-18, Tumor necrosis factor (TNF)-a , Tumor necrosis factor receptor two (TNF-RII) | Preoperative (1-2 days preoperative) and 3-4 days postoperative and 6 weeks postoperative and 12 weeks postoperative
  Change in serum levels of cytokines (Interleukin (IL)-6 , IL-10, IL-18, Tumor necrosis factor (TNF)-a , Tumor necrosis factor receptor two (TNF-RII)

CONTACTS AND LOCATIONS:
Overall Officials: Eliska Potlukova, PhD, Principal Investigator — Klinik für Innere Medizin, Universitätsspital Basel
Locations (1):
- University Hospital Basel, Basel, Switzerland